CLINICAL TRIAL: NCT01308346
Title: ABSORB PHYSIOLOGY Clinical Investigation: Clinical Evaluation of the Short and Long-Term Effects of the Abbott Vascular Everolimus-Eluting Bioresorbable Vascular Scaffold on Coronary Artery Blood Flow and Physiological Responsiveness
Brief Title: ABSORB PHYSIOLOGY Clinical Investigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a challenging protocol inclusion/ exclusion criteria, only one subject was enrolled since the trial was initiated in June 2011.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 10-390
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease
Keywords: Bioabsorbable; Coronary Stent; Everolimus; drug eluting stents; stents; angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioresorbable Vascular Scaffold (BVS) (Experimental): Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS)
  Interventions: Device: Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS)
- XIENCE V® or XIENCE PRIME® (Active Comparator): XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) or XIENCE PRIME®
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent System (EECSS)

INTERVENTIONS:
Device: Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS) — Bioabsorbable Everolimus Eluting Coronary Stent
  Arms: Bioresorbable Vascular Scaffold (BVS)
Device: XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) — XIENCE V® Everolimus Eluting Coronary Stent System (EECSS)
  Arms: XIENCE V® or XIENCE PRIME®

SUMMARY:
The target enrollment goal for the trial was to enroll 36 subjects. However due to a challenging protocol inclusion/ exclusion criteria, only one subject was enrolled since the trial was initiated in June 2011.

To evaluate the following in participants undergoing coronary artery scaffolding/stenting for significant coronary artery disease:

* The acute (post-implantation) effect of an implanted bioresorbable vascular scaffold (BVS) or metallic drug eluting stent (mDES) on coronary blood flow and physiological responsiveness of the target coronary artery
* The long-term (2 years) effect of an implanted BVS or mDES on coronary blood flow and physiological responsiveness of the target coronary artery

DETAILED DESCRIPTION:
* Prospective, randomized, single-blinded, multi-center clinical investigation comparing target vessel and non-intervened, self-control vessel within participants and between participants undergoing BVS or mDES deployment for the treatment of a single de novo native coronary artery lesion
* The investigation will include two arms:

  * Study device (BVS) arm: Abbott Vascular's Everolimus-Eluting Bioresorbable Vascular Scaffold
  * Control device (mDES) arm: Abbott Vascular's Everolimus-Eluting XIENCE V or XIENCE PRIME

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be a male of at least 18 years of age or a female that is post-menopausal and not on hormone replacement therapy.
2. Participant is able to verbally confirm understanding of risks, benefits and treatment alternatives and he/she or his/her legally authorized representative must provide written informed consent prior to any clinical investigation related procedure, as approved by the appropriate Ethics Committee of the respective clinical site.
3. Participant must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia with a positive functional study).
4. Participant must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Participant must agree to undergo all clinical investigation plan-required follow-up visits.
6. Participant must agree not to participate in any other clinical investigation for a period of 2 years following the index procedure. This includes clinical trials of medications and invasive procedures. Only questionnaire-based studies are allowed.

Angiographic Inclusion Criteria:

1. A single de novo native coronary artery lesion suitable to be treated by either a BVS or a mDES.
2. Target lesion must be located in a native coronary artery in which the mean proximal and distal vessel diameter of the target lesion (Dmean) fall within the range of ≥ 2.25 mm and ≤ 3.25 mm and the target lesion length measures ≤ 22 mm as assessed by IVUS.
3. Target lesion must be located in the main branch of a major epicardial vessel (i.e., LAD, LCX, or RCA) with a visually estimated diameter stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 1.
4. Participant must have an additional angiographically smooth (< 40% diameter stenosis) non-target vessel to act as an intra-participant control vessel (self-control vessel). The self-control vessel must be the main branch of a major epicardial vessel (i.e., LAD, LCX, or RCA).
5. Coronary anatomy must be suitable for IVUS, OCT, and pressure and flow wire instrumentation.

General Exclusion Criteria:

1. Participant has a known diagnosis of spontaneous acute myocardial infarction (AMI) within 14 days preceding the index procedure.
2. Participant has high-risk acute coronary syndrome (e.g., dynamic ST-T wave change on ECG or recurrent chest pain/nitrate-unresponsive prolonged chest pain at rest within 48 hours prior to the index procedure).
3. Participant has any evidence of myocardial infarct in the territory subtended by the proposed target vessel or self-control vessel.
4. Participant has current unstable arrhythmias.
5. Participant has chronic atrial fibrillation.
6. Participant has a known left ventricular ejection fraction (LVEF) < 40%.
7. Participant has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant.
8. Participant has previously had CABG or mitral or aortic valve repair/replacement.
9. Participant is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the index procedure.
10. Participant is receiving immunosuppressant therapy or has known immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.).
11. Participant has a chronic systemic condition or medication likely to interfere with coronary physiology and/or conduit artery function (e.g., chronic inflammatory condition, chronic renal failure, or chronic obstructive pulmonary disease).
12. Participant has known renal insufficiency.
13. Participant is receiving or scheduled to receive any planned radiotherapy.
14. Participant is receiving chronic anticoagulation therapy (e.g., heparin, coumadin) at the onset of the clinical investigation.
15. Participant has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, anti-platelet medications specified for use in the study (clopidogrel, prasugrel and ticlopidine, inclusive), everolimus, poly (L-lactide), poly (DL-lactide), cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers, or contrast sensitivity that cannot be adequately pre-medicated.
16. Elective surgery is planned within the first 6 months after the index procedure that will require discontinuing aspirin, clopidogrel, prasugrel, or ticlopidine.
17. Participant has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis) within 7 days prior to the index procedure.
18. Participant has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
19. Participant has had a cerebrovascular accident/stroke (CVA) or transient ischemic neurological attack (TIA) within the past 6 months.
20. Participant has had a significant gastro-intestinal or significant urinary bleed within the past 6 months.
21. Participant has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.
22. Participant has a history of paradoxical exercise-induced vasoconstriction that is consistent with myocardial bridging in the coronary anatomy.
23. Participant has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that in the judgment of the Investigator may cause non-compliance with the clinical investigation plan, confound the data interpretation or is associated with a limited life expectancy.
24. Participant is currently participating in another clinical investigation that has not yet reached its primary endpoint.
25. Percutaneous interventions for lesions in the third major epicardial vessel (the one that does not contain the target or the self-control vessel) were performed within 30 days preceding the index procedure or are planned to be done within 6 months following the index procedure.
26. Planned PCI procedures in the target vessel (and/or any of its side branches) or the self-control vessel (and/or any of its side branches) within 2 years following the index procedure.
27. Participant who does not suspend drugs that will influence vaso-function.

Angiographic Exclusion Criteria

1. Target lesion meets any of the following criteria:

   1. Left main location;
   2. RCA aorto-ostial location (within 10 mm from expected proximal stent/scaffold edge);
   3. LAD or LCX ostial location (within 10 mm from expected proximal stent/scaffold edge);
   4. Involves a bifurcation with a side branch ≥ 2 mm in diameter, an ostial lesion > 40% stenosed by visual estimation, or a side branch requiring pre-dilatation;
   5. Total occlusion (TIMI flow 0) prior to wire crossing;
   6. Excessive tortuosity proximal to or within the lesion;
   7. Extreme angulation (≥ 90°) proximal to or within the lesion;
   8. Heavy calcification in the lesion;
   9. Located in a side branch.
2. Participant has a high probability that a procedure other than pre-dilatation, scaffold/stent implantation, and post-dilatation (if applicable) will be required at the time of index procedure for treatment of the target vessel (e.g., atherectomy, cutting balloon or brachytherapy).
3. The target vessel (and/or any of its side branches) or the self-control vessel (and/or any of its side branches) contains visible thrombus.
4. The target vessel or the self-control vessel has previously been treated by any PCI procedures.
5. A side branch of the target vessel or a side branch of the self-control vessel has received any percutaneous interventions within 30 days prior to the index procedure.
6. Another clinically significant lesion is located in the target vessel (and/or any of its side branches) or the self-control vessel (and/or any of its side branches) that may require PCI treatments within 2 years following the index procedure.
7. Participant has evidence of myocardial bridging in the coronary anatomy during the angiographic evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Coronary artery endothelial responsiveness | Post procedure
  Change of vessel diameter by 1) pacing, 2) hand-grip and 3) acetylcholine injection

SECONDARY OUTCOMES:
Coronary artery cross-sectional compliance and cross-sectional distensibility | Post procedure
  Cross-sectional compliance is defined as change in area per unit change in pressure; cross-sectional distensibility is defined as compliance/diastolic cross-sectional area.
Target artery endothelial shear stress distribution | Post procedure
  Wall Shear Stress (WSS) will be determined from flow velocity and blood viscosity
Wave intensity patterns in the coronary arteries | Post procedure
  Looking at re-distribution of energy in the blood flow along the coronary artery.
Systolic and diastolic coronary artery impedance | Post procedure
Clinical device success | Post procedure
  Successful delivery and deployment of the Clinical Investigation scaffold at the target lesion and successful withdrawal of the scaffold delivery system.
Clinical Procedure Success | during the hospital stay with a maximum of 7 days post index procedure.
  Successful delivery and deployment of the Clinical Investigation scaffold at the target lesion and successful withdrawal of the scaffold delivery system without the occurrence of ischemia driven major adverse cardiac event (MACE).
Cardiac Death (CD) | 180 days
Cardiac Death (CD) | 1 year
Cardiac Death (CD) | 2 years
Myocardial Infarction (MI) | 180 days
Myocardial Infarction (MI) | 1 year
Myocardial Infarction (MI) | 2 years
Target Vessel Myocardial Infarction (TV-MI) | 180 days
Target Vessel Myocardial Infarction (TV-MI) | 1 year
Target Vessel Myocardial Infarction (TV-MI) | 2 years
All Death, All MI, All Revascularization (DMR) | 180 days
All Death, All MI, All Revascularization (DMR) | 1 year
All Death, All MI, All Revascularization (DMR) | 2 years
Ischemia-Driven MACE (ID-MACE) | 180 days
Ischemia-Driven MACE (ID-MACE) | 1 year
Ischemia-Driven MACE (ID-MACE) | 2 years
Ischemia-Driven Target Vessel Failure (ID-TVF) | 180 days
Ischemia-Driven Target Vessel Failure (ID-TVF) | 1 year
Ischemia-Driven Target Vessel Failure (ID-TVF) | 2 years
Ischemia-Driven Target Vessel Revascularization (ID-TVR) | 180 days
Ischemia-Driven Target Vessel Revascularization (ID-TVR) | 1 year
Ischemia-Driven Target Vessel Revascularization (ID-TVR) | 2 years
Ischemia-Driven Self-Control Vessel Revascularization (ID-SCVR) | 180 days
Ischemia-Driven Self-Control Vessel Revascularization (ID-SCVR) | 1 year
Ischemia-Driven Self-Control Vessel Revascularization (ID-SCVR) | 2 years
Ischemia-Driven Non-Target, Non-Self-Control Vessel Revascularization (ID-NTNSCVR) | 180 days
Ischemia-Driven Non-Target, Non-Self-Control Vessel Revascularization (ID-NTNSCVR) | 1 year
Ischemia-Driven Non-Target, Non-Self-Control Vessel Revascularization (ID-NTNSCVR) | 2 years
Ischemia-Driven Target Lesion Revascularization (ID-TLR) | 180 days
Ischemia-Driven Target Lesion Revascularization (ID-TLR) | 1 year
Ischemia-Driven Target Lesion Revascularization (ID-TLR) | 2 years
Scaffold/Stent thrombosis | 180 days
Scaffold/Stent thrombosis | 1 year
Scaffold/Stent thrombosis | 2 years
Coronary artery endothelial responsiveness | 2 years
  Change of vessel diameter by 1) pacing, 2) hand-grip and 3) acetylcholine injection
Coronary artery cross-sectional compliance and cross-sectional distensibility | 2 years
  Cross-sectional compliance is defined as change in area per unit change in pressure; cross-sectional distensibility is defined as compliance/diastolic cross-sectional area.
Target artery endothelial shear stress distribution | 2 years
  Wall Shear Stress (WSS) will be determined from flow velocity and blood viscosity
Wave intensity patterns in the coronary arteries | 2 years
  Looking at re-distribution of energy in the blood flow along the coronary artery.
Systolic and diastolic coronary artery impedance | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Meredith, Prof, MD, Principal Investigator — Monash Medical Center; James Cameron, Prof, MD, Principal Investigator — Monash Medical Center
Locations (6):
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Monash Medical Centre, Melbourne
- Queen Elizabeth, Hong Kong, China
- Maasstad Ziekenhuis, Rotterdam, Netherlands
- National Heart Centre Singapore, Singapore, Singapore